CLINICAL TRIAL: NCT03307486
Title: Fetal and Maternal Repercussions of Gestational Diabetes After the Adoption of the Diagnostic Criteria Proposed by the International Association of Diabetes and Pregnancy Study Groups (IADPSG): a Cohort Study
Brief Title: Gestational Diabetes: a Cohort Study
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 48868915.9.0000.0068
Record Dates: First submitted 2017-07-25; First posted 2017-10-11 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-07

CONDITIONS: Gestational Diabetes; Diabetes, Gestational; Diabetes Mellitus in Pregnancy; Diabetes Mellitus, Type 2
Keywords: Gestational diabetes; Type 2 DM after GDM
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gestational diabetes: Women diagnosed with GDM according to the IADPSG criteria, either by abnormal fasting plasma glucose or by abnormal oral glucose tolerance test.

SUMMARY:
Gestational diabetes (GDM) is the most common hormonal complication during pregnancy. Its occurrence implies an increased risk of maternal and fetal complications and, therefore, its diagnosis and treatment are extremely important. Since the adoption of the new diagnostic criteria proposed by the International Association of Diabetes and Pregnancy Study Groups (IADPSG) in 2010, an increasing number of cases of mild hyperglycemia have demanded follow-up and treatment. The need and benefit of treatment in these cases of mild hyperglycemia has been discussed worldwide. Women who have been diagnosed with GDM are at increased risk for type 2 DM in the years following gestation. Other factors (such as lipid profile, obesity, adipokine dosage) may also be related to the repercussions of GDM on the maternal-fetal binomial, since gestations with satisfactory glycemic control can also present complications related to the disease and increased risk of type 2 DM in the long term. The present study aims to investigate factors associated with the need for insulin use, the occurrence of perinatal complications, nutritional status, physical activity and weight retention one year after delivery and the postpartum diagnosis of type 2 DM 10 years after delivery in women diagnosed with GDM according to the current criteria suggested by the IADPSG.

ELIGIBILITY:
Inclusion Criteria:

* single pregnancies
* absence of glucose intolerance prior to gestation (defined by prior diagnosis of polycystic ovarian syndrome or fasting glycemia ≥100mg / dl or 2hr post-overload with 75g glucose ≥ 140mg / dL or glycated hemoglobin ≥ 5.7% previously to pregnancy)
* absence of chronic use of glucocorticoids or antiretroviral drugs for HIV virus, given its diabetogenic effect and potential confounding
* diagnosis of GDM according to diagnostic criteria proposed by the IADPSG, namely: initial fasting blood glucose ≥ 92mg / dL OR oral glucose tolerance test of 75g with fasting ≥ 92mg / dL or after1h ≥ 180mg / dL or after 2h ≥ 153mg / dL
* Agreement with the informed consent term for patients who will be followed prospectively
* Agreement with the free and informed consent term for recall and reassessment of the patients identified in the retrospective analysis of the data

Exclusion Criteria:

* loss to follow up during pregnancy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were diagnosed with gestational diabetes after the adoption of the diagnostic criteria proposed by the IADPSG (June 2011) will be evaluated retrospectively and prospectively in the high-risk prenatal outpatient clinic of the Obstetric Clinic of the Hospital das Clínicas of the Medical School of the University of São Paulo (HCFMUSP), a tertiary teaching hospital in Sao Paulo, Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2015-09-17 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of type 2 DM after GDM | 10 years
  To evaluate clinical, nutritional and laboratory factors as tools to predict the diagnosis of type 2 DM, carbohydrate intolerance or postpartum metabolic syndrome in women who had GDM

SECONDARY OUTCOMES:
Need of insulin | during pregnancy
  To evaluate clinical and laboratory factors as tools to predict the need of insulin during pregnancy
Weight at birth | during pregnancy and delivery
  To evaluate clinical, ultrasonographic and laboratory factors as tools to predict weight at birth (grams)
Route of delivery | during pregnancy and delivery
  To evaluate clinical, ultrasonographic and laboratory factors as tools to predict the route of delivery
Neonatal Hypoglycemia | during pregnancy and delivery
  To evaluate clinical, ultrasonographic and laboratory factors as tools to predict neonatal hypoglycemia
Obesity in the offspring | 10 years
  To evaluate clinical, ultrasonographic and laboratory factors as tools to predict obesity in the offspring of women with GDM
Hypertension in the offspring | 10 years
  To evaluate clinical, ultrasonographic and laboratory factors as tools to predict hypertension in the offspring of women with GDM
Body composition | during pregnancy, 6 months postpartum and one year after delivery
  To assess the body composition of women with gestational diabetes during pregnancy, 6 months postpartum and one year postpartum
Physical activity | during pregnancy , 6 months postpartum and 1 year after delivery
  identify the level of daily physical activity of women with gestational diabetes during pregnancy, 6 months postpartum and one year postpartum
Eating habits | during pregnancy, 6 months postpartum and 1 year after delivery
  to verify the eating habits of women with gestational diabetes during pregnancy, 6 months postpartum and one year postpartum
Weight retention | during pregnancy, 6 months postpartum and 1 year after delivery
  To study association between levels of physical activity and dietary intake and the weight retention in women with gestational diabetes during pregnancy, 6 months postpartum and one year postpartum
Route of delivery vs physical activity | during pregnancy and delivery
  to study association between the level of physical activity in women with gestational diabetes during pregnancy and the route of delivery (cesarian or vaginal birth)
Route of delivery vs eating habits | during pregnancy and delivery
  to study association between the eating habits in women with gestational diabetes during pregnancy and the route of delivery (cesarian or vaginal birth)
Fetal weight at birth vs physical activity | during pregnancy and delivery
  to study association between physical activity in women with gestational diabetes during pregnancy and the fetal weight at delivery (grams)
Fetal weight at birth vs eating habits | during pregnancy and delivery
  to study association between eating habits in women with gestational diabetes during pregnancy and the fetal weight at delivery (grams)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil